CLINICAL TRIAL: NCT00317538
Title: Open-label, Pilot Protocol of Patients With Rheumatoid Arthritis Who Switch to Infliximab After Incomplete Response to Etanercept
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor Ortho Biotech Services, L.L.C. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR003136; NCT00094471 (obsolete NCT alias)
Record Dates: First submitted 2006-04-21; First posted 2006-04-25 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Switching; Structural Damage; MRI
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab; Etanercept

INTERVENTIONS:
Drug: infliximab, etanercept

SUMMARY:
The purpose of this study, in patients with rheumatoid arthritis who have had an incomplete response to etanercept and methotrexate (MTX), are to evaluate: safety and evidence of therapeutic benefit of infliximab and methotrexate, the levels (pharmacokinetics) of etanercept and infliximab and antibodies (immunogenicity) to etanercept and infliximab in patients blood, whether switching from etanercept to infliximab changes progression of structural damage over the study period, and whether specific markers in the blood (pharmacodynamics) correlate with therapeutic response or benefit.

DETAILED DESCRIPTION:
Therapeutic agents designed to bind and block the biological activities of tumor necrosis factor-alpha (TNFa) have been shown to be effective in the treatment of rheumatoid arthritis (RA). Two anti-TNFa agents are currently marketed for the treatment of RA; etanercept (Enbrel®) and infliximab (REMICADE®). Clinical trials have shown that both of these agents rapidly improve signs and symptoms associated with RA in the majority of patients. Moreover, they slow, and may even arrest or improve, the joint structural damage that accompanies RA.

While infliximab and etanercept are designed to block the biological activities of TNFa, these agents are sufficiently different in their structure that they may have distinct, as well as overlapping, mechanisms of action. The clearest evidence of this possibility can be inferred from their differential activities in certain diseases such as Crohn's disease in which infliximab, but not etanercept, shows beneficial therapeutic activity. The mechanism of their differential biological activities is not known. That infliximab and etanercept show differential activities in other diseases suggests that they may also have distinct effects in RA.

The question of whether or not patients who fail to respond to or incompletely respond to etanercept can still respond to infliximab has potentially important therapeutic implications. Evidence that such patients respond to infliximab could support the notion that these agents have important differences in their mechanisms of action, or could be explained by the presence of antibodies to etanercept. More importantly, it would suggest that therapeutic failure of one TNFa-blocker does not necessarily predict failure of all TNFa-targeting agents. Such a finding could open important therapeutic alternatives to RA patients and is of clear importance because this class of biologics (biologic agent) represents the most significant advance to date in the treatment of RA.

This initial open-label, pilot study will be performed in approximately 24 patients with RA who have who have achieved some therapeutic benefit from treatment with concomitant etanercept and MTX for a minimum of 3 months, but the response must be an incomplete response, and patients must have a minimum of 9 tender and 6 swollen joints while receiving concomitant etanercept and MTX. It will assess safety and evidence of therapeutic benefit of infliximab in this patient population. The study will examine any differences in the pharmacokinetics and immunogenicity of etanercept and infliximab in patients who are incomplete responders to etanercept.

This is an open-label, exploratory study and no formal hypothesis is being tested. This study will provide a preliminary assessment of safety and evidence of therapeutic benefit of infliximab plus MTX in patients with RA who are incomplete responders to etanercept plus MTX. One group will receive intravenous infliximab infusions at a dose of 3 mg/kg at weeks 0, 2, 6 14 and 22. The second group will receive etanercept injections, 25 mg subcutaneously twice weekly from week 0 through 16 and may receive intravenous infliximab infusions at 3 mg/kg on weeks 16, 18 & 22.

ELIGIBILITY:
Inclusion Criteria:

* Patients have a diagnosis of RA according to the revised 1987 criteria of the American Rheumatism Association
* Have been receiving background MTX for at least 2 months prior to week -4
* Have been receiving a stable etanercept dose of 25 mg subcutaneously twice weekly for at least 2 months prior to week -4
* Must have been using oral or parenteral MTX for the 2 months prior to screening and at a stable dose of 7.5 to 25 mg per week between week -4 and week 0
* Have shown improvement in signs and symptoms of RA in response to etanercept and MTX according to both the patient and the treating physician
* Have active disease as defined by both a TJC of at least 9 (on the 68 joint set) and SJC of at least 6 (on the 66 joint set)
* Have a documented negative reaction to a purified protein derivative (PPD) skin test (PPD induration< 5 mm) performed within 3 months prior to the week 0 visit

Exclusion Criteria:

* Patients have been receiving corticosteroids (ie, via any route) at doses > 10 mg prednisone equivalent daily or have not been taking a stable dose of corticosteroids for at least 1 month prior to week -4
* Have started receiving nonsteroidal anti-inflammatory drugs (NSAIDs) within 1 month of week -4 or have not been on a stable dose of NSAIDs for at least 1 month prior to week -4
* Have received disease modifying anti-rheumatic drugs (DMARDs) or immunosuppressives (except MTX) for at least 1 month prior to week 0

Patients who have received any prior treatment with infliximab or with any other therapeutic agent targeted at reducing TNF, except etanercept, (e.g.pentoxifylline or thalidomide)

* Patients with a concomitant diagnosis of Congestive Heart Failure, including medically controlled asymptomatic patients
* Any current known malignancy or history of malignancy within the previous 5 years
* Serious infection within the past 3 months or history of chronic infection such as hepatitis, pneumonia, or pyelonephritis in the previous 3 months, any opportunistic infections
* known substance abuse (drug or alcohol) within the previous 3 years
* Are pregnant, nursing, or planning pregnancy (both men and women) during the trial or within the 6-month period thereafter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2003-06; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Evaluate safety and evidence of therapeutic benefit of infliximab and methotrexate, in patients with rheumatoid arthritis who have had an incomplete response to etanercept and methotrexate (MTX), at week 16

SECONDARY OUTCOMES:
Evaluate pharmacokinetics, immunogenicity, structural damage and pharmacodynamics over the study period

CONTACTS AND LOCATIONS:
Overall Officials: Centocor Ortho Biotech Services, L.L.C. Clinical Trial, Study Director — Centocor Ortho Biotech Services, L.L.C.

REFERENCES:
- See also: Open-label, Pilot Protocol of Patients with Rheumatoid Arthritis Who Switch to Infliximab after Incomplete Response to Etanercept — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=129&filename=CR003136_CSR.pdf